CLINICAL TRIAL: NCT06556342
Title: Efficacy and Safety of FRD001 Injection in Ultrasound Contrast Imaging for the Differential Diagnosis of Benign and Malignant Ovarian Masses in Women
Brief Title: The Efficacy and Safety of FRD001 in Ultrasound Contrast Imaging for Malignant Ovarian Masses in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-TJ-FRDOC
Record Dates: First submitted 2024-08-11; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic cohort (Experimental): This trial will adopt a self-controlled design, where each participant will first undergo gray-scale/power Doppler ultrasound imaging, followed by FRD001 injection-enhanced ultrasound imaging. At least 198 subjects will be needed, which includes 79 participants with malignant tumors (N1) and 119 with benign conditions (N2). All screening assessments for each participant will be conducted within 7 days prior to the administration of the investigational medicinal product (IMP), including the day of administration. Safety observations will continue for 72 ± 24 hours post-IMP administration. Pathological results for the target lesions will be collected within 30 days following the IMP imaging examination.
  Interventions: Drug: FRD001

INTERVENTIONS:
Drug: FRD001 — FRD001 injection is a lipid-based second-generation ultrasound contrast agent. FRD001 injection in ultrasound contrast imaging could enhance the differentiation between benign and malignant ovarian masses in women, using gray-scale and power Doppler ultrasound as controls.

SUMMARY:
This is a Prospective, Self-Controlled, Open-Label, Multicenter Clinical Trial. The purpose of this study is to demonstrate the efficacy and safety of FRD001 injection in ultrasound contrast imaging for the differentiation between benign and malignant ovarian masses in women, using gray-scale and power Doppler ultrasound as controls. This trial will adopt a self-controlled design, where each participant will first undergo gray-scale/power Doppler ultrasound imaging, followed by FRD001 injection-enhanced ultrasound imaging. The target population is assumed to have a malignancy prevalence (P) of 40%, with an expected sensitivity of gray-scale/power Doppler ultrasound at 70%. It is hypothesized that the sensitivity of FRD001 injection-enhanced ultrasound will improve by 20%, reaching an anticipated sensitivity of 90%. The significance level (α) is set at 0.05, with a power (1-β) of 80%, and an inconsistency ratio (D) of 0.34. Based on these parameters, a total sample size (N) of 178 cases is required. Considering a 10% dropout rate, at least 198 subjects will be needed, which includes 79 participants with malignant tumors (N1) and 119 with benign conditions (N2). All screening assessments for each participant will be conducted within 7 days prior to the administration of the investigational medicinal product (IMP), including the day of administration. Safety observations will continue for 72 ± 24 hours post-IMP administration. Pathological results for the target lesions will be collected within 30 days following the IMP imaging examination. The efficacy of the IMP in differentiating between benign and malignant ovarian masses will be evaluated against pathological results, which will serve as the gold standard. This comprehensive approach will provide crucial insights into the diagnostic capabilities of FRD001 injection, potentially enhancing clinical decision-making in the management of ovarian masses.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet the following inclusion criteria to be eligible for enrollment in this study:

* Female participants aged 18 to 75 years (inclusive of the age limits);
* Patients with untreated unilateral or bilateral, unilocular or multilocular cystic/solid masses;
* Expected survival of at least 3 months;
* ECOG performance status of 0 to 2 for participants with malignant tumors;
* Organ function levels must meet the following requirements: a. Hematology: WBC ≥ 3 × 10^9/L, ANC ≥ 1.5 × 10^9/L, Hb ≥ 90 g/L, PLT ≥ 75 × 10^9/L; b. Liver function: TBIL ≤ 1.5 × ULN, ALT and AST ≤ 3 × ULN (≤ 5 × ULN for patients with liver metastases); c. Kidney function: Cr ≤ 1.5 × ULN; d. Coagulation function: Prothrombin time (PT) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, International normalized ratio (INR) ≤ 1.5 × ULN; e. Electrolytes: Corrected magnesium ≥ LLN, with allowance for correction of electrolytes during screening; f. Cardiac function: Left ventricular ejection fraction ≥ 50%; g. Pulse oximetry ≥ 93%;
* Women of childbearing potential must use effective contraception during the study (effective contraceptive methods include sterilization, intrauterine hormonal devices, condoms, contraceptive pills/devices, abstinence, or vasectomy);
* Participants must fully understand the purpose, nature, methods, and potential adverse reactions of the trial, voluntarily agree to participate, and sign a written informed consent form, demonstrating the ability to adhere to the protocol requirements to complete the study.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for enrollment:

* Patients with benign teratomas;
* Patients who have undergone total removal of the uterine appendages;
* Patients with congenital malformations of the reproductive system;
* Patients who have received radiotherapy, chemotherapy, or invasive procedures (including but not limited to radiofrequency ablation) during the administration of the investigational medicinal product (IMP) and the confirmatory diagnostic examination;
* Women planning to become pregnant within 6 months, currently pregnant, or breastfeeding, or women of childbearing potential with a positive pregnancy test during the screening period;
* Individuals allergic to the components of FRD001 injection or with a history of other severe allergies;
* Insufficient acoustic window indicated by ultrasound examination during screening or prior examinations;
* Presence of contraindications for imaging examinations related to the study protocol;
* Conditions such as adult respiratory distress syndrome, severe emphysema, pulmonary vasculitis, or pulmonary embolism;
* Severe cardiovascular or cerebrovascular diseases, including but not limited to: a. Significant cardiac rhythm or conduction abnormalities that require clinical intervention, such as ventricular arrhythmias, second- to third-degree atrioventricular block, or QTc interval ≥ 450 ms; b. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other cardiovascular events of grade 3 or higher within 6 months prior to the first dose; c. New York Heart Association (NYHA) functional classification ≥ II or left ventricular ejection fraction (LVEF) < 50%;
* Known severe pulmonary hypertension or uncontrolled systemic hypertension; uncontrolled hypertension (for individuals <60 years old, systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg; for individuals ≥ 60 years old, systolic blood pressure ≥ 150 mmHg and diastolic blood pressure ≥ 90 mmHg);
* Patients with symptomatic brain metastases requiring treatment;
* Individuals with severe or uncontrolled mental illness;
* Presence of active infections requiring systemic treatment or uncontrolled infections within 14 days prior to starting the investigational drug;
* Positive tests for antibodies to human immunodeficiency virus (HIV), hepatitis C virus (HCV), or Treponema pallidum; positive hepatitis B virus (HBV) surface antigen;
* History of right-to-left, bidirectional, or transient right-to-left cardiac shunts;
* History of alcohol or drug abuse/dependence;
* Participation in other clinical trials involving investigational drugs within 30 days prior to screening;
* Any medications or treatments deemed by the investigator to potentially interfere with trial data or cause severe side effects that have not been fully washed out prior to enrollment;
* Any other conditions deemed inappropriate for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with ovarian mass.
Enrollment: 198 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 years
  The primary endpoint is sensitivity, calculated using pathological results as the gold standard, according to the previously established formulas.

SECONDARY OUTCOMES:
Specificity | 1 years
  The secondary endpoints include specificity, calculated using pathological results as the gold standard, according to the previously established formulas.
Adverse events (AE) and serious adverse events (SAE) | 1 years
  Adverse events (AE) and serious adverse events (SAE) are assessed according to the common terminology criteria for adverse events (NCI-CTCAE) version 5.0. All adverse events occurring in subjects during the clinical trial are observed, and their clinical characteristics, severity, occurrence time, resolution time, management measures, and outcomes are recorded, along with an assessment of their correlation with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No